CLINICAL TRIAL: NCT06618508
Title: Comparison of Efficacy and Safety Between Manual Debridement and Phototherapeutic Keratectomy (PTK) in the Treatment of Corneal Basement Membrane Dystrophy
Brief Title: Manual Debridement Vs Phototherapeutic Keratectomy in the Treatment of Corneal Basement Membrane Dystrophy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Samir Jabbour, Dr Samir Jabbour, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-12106
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Epithelial Basement Membrane Dystrophy
MeSH Terms: conditions — Corneal dystrophy, epithelial basement membrane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual debridement (Active Comparator): Manual debridement is a technique that has existed since 1952 and whose objective is to remove the irregular epithelium by scraping with an instrument, thus allowing the formation of a new superficial layer. Some surgeons use 20% ethanol which they apply to the cornea to debride it before using a blade or sponge to complete the procedure. In this technique, the basement membrane is preserved. This method is still used being simple and cost effective. Its effectiveness in the treatment of recurrent corneal erosions is demonstrated by a success rate estimated at 85%. Thus, it is one of the methods of treating epithelial basement membrane dystrophy. However, the recurrence rate associated with manual debridement is up to 24%, and the average duration before a first recurrence is estimated at 6 months. The formation of corneal opacities was recorded between 7 and 41 days following the intervention.
  Interventions: Procedure: Manual debridement
- Phototherapeutic keratectomy (Experimental): Over the past two decades, phototherapeutic keratectomy (PTK) has become an increasingly used approach for the treatment of several anterior corneal pathologies, including epithelial basement membrane dystrophy. This technique consists of directing a 193nm excimer laser towards the epithelial surface in order to break the molecular bonds between cells. PTK appears to be a more reliable, safe and precise alternative to manual debridement. Unlike manual debridement, PTK completely obliterates the basement membrane which would promote a reduction in the recurrence rate according to some experts. Thus, the success rate without recurrence has been estimated between 46 to 100% by certain studies and the associated complications are minimal.
  Interventions: Procedure: Phototherapeutic keratectomy

INTERVENTIONS:
Procedure: Manual debridement — Traditional technique which consists of scraping off the irregular epithelium to allow a new layer to form.
  Arms: Manual debridement
Procedure: Phototherapeutic keratectomy — New technique which has been increasingly used and which consists of a 193nm excimer laser that breaks molecular bonds between cells on the epithelial surface.
  Arms: Phototherapeutic keratectomy

SUMMARY:
Of the few comparisons made in the existing literature, the results of PTK are comparable to those documented for manual debridement (MD). However, the shorter length of follow-up in patients with MD may have underestimated the associated complications. Our study, therefore, aims to offer a comparison between these two techniques to clarify the choice of effective treatment with a good safety profile.

DETAILED DESCRIPTION:
Epithelial Basement Membrane Dystrophy (EBMD) affects the anterior cornea, impacting about 2% of the population. EBMD is characterized by alterations and duplications of the basement membrane, a tissue layer that connects the epithelium to the underlying eye tissue. Dysfunction of the basement membrane prevents proper adhesion of the overlying epithelium, leading to recurrent corneal erosions. Additionally, tissue protrusions infiltrate the epithelium, creating surface irregularities that cause symptoms like blurred vision and irregular corneal topographies. This abnormal proliferation results in microcysts and corneal irregularities resembling fingerprints and maps. These surface irregularities can be observed in optical coherence tomography (OCT) images showing epithelial thickening. Non-invasive medical treatments are the first line of therapy, including lubricating drops and hypertonic solutions to protect the ocular surface and promote epithelial adhesion. For corneal erosions, soft contact lenses are used to aid healing. Surgical interventions such as manual debridement and phototherapeutic keratectomy (PTK) are required in refractory cases. These are also indicated for patients preparing for cataract surgery to optimize preoperative corneal measurements and postoperative optical outcomes. Manual debridement (MD), a technique since 1952, involves scraping off the irregular epithelium to allow a new layer to form. Some surgeons use 20% ethanol on the cornea before scraping with a blade or sponge, preserving the basement membrane. This method is simple, cost-effective, and has an 85% success rate in treating recurrent corneal erosions. However, recurrence rates are up to 24%, with the first recurrence typically within six months. Corneal opacities can form between 7 and 41 days post-procedure. Over the past two decades, PTK has become increasingly used for anterior corneal pathologies, including EBMD. PTK uses a 193nm excimer laser to break molecular bonds between cells on the epithelial surface. It is considered a more reliable, safe, and precise alternative to manual debridement, completely obliterating the basement membrane and potentially reducing recurrence rates. Success rates without recurrence range from 46% to 100%, with minimal complications. Unlike manual debridement, PTK may induce a hyperopic shift, which stabilizes within a year. Corneal erosions and pain recur at about 13% over an average of 9.7 months. Comparative studies between these two methods are scarce, and more data is needed to favor one technique over the other. Limited comparisons suggest PTK results are comparable to manual debridement, though shorter follow-ups in MD patients may underestimate associated complications. Our study aims to compare these techniques to describe the efficacy and safety of both treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Ability to give free and informed consent
* At least 1-year follow-up possible
* Patients with bilateral basal membrane corneal dystrophy who are symptomatic (recurrent corneal erosions, visual disturbances) and are candidates for bilateral surgery.

Exclusion Criteria:

* Patient under 18 years of age;
* History of ocular infection with herpes simplex virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of corneal basement membrane dystrophy | Day 1, week 1 and months 1, 3, 6, 12 and 24 months
  Evaluated with slit-lamp morphological findings (maps, "fingerprint" lines, epithelial microcysts), imaging results including OCT (thickened basement membrane and epithelial irregularities) and patient symptoms (redness, pain, photophobia, associated with erosions).

SECONDARY OUTCOMES:
Corneal haze formation assessed by a corneal haze gradation scale | 1, 3, 6, 12 and 24 months
  0: Clear with no opacity seen by any method of microscopic slit-lamp examination.
  0.5: Trace or faint haze seen only by indirect, broad tangential illumination.
  1. Haze of minimal density seen with difficulty with direct or diffuse examination.
  2. Mild haze easily visible with direct focal slit lamp illumination.
  3. Moderate opacity that partially obscured details of iris.
  4. Severe opacity that completely obscured the details of intraocular structures.
Contrast sensitivity with the CSV-1000 Contrast Sensitivity chart with glare | 1,3,6,12 and 24 months
  Standardized contrast sensitivity test.
Patient comfort using the Wong-Baker FACES pain scale | Day 1, week 1, month 1, month 3, month 6 and month 12
  0 = no hurt; 2= hurts a little bit; 4=hurts little more; 6=hurts even more; 8=hurts whole lot; 10=hurts worst
Post-operative complications | Day 1, week 1, month 1, month 3, month 6 and month 12
  Post-operative complications include persistent epithelial deficits, formation of subepithelial corneal opacities, infectious keratitis, reactivation of herpes simplex virus, scarring, and corneal infiltrates.
Best corrected distance visual acuity (BCVA) | 1,3,6,12 and 24 months
  This is the visual acuity measured using an eye chart. To achieve best possible visual acuity, corrective lenses are used.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jabbour, MD,CM,FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee WS, Lam CK, Manche EE. Phototherapeutic keratectomy for epithelial basement membrane dystrophy. Clin Ophthalmol. 2016 Dec 16;11:15-22. doi: 10.2147/OPTH.S122870. eCollection 2017. PMID 28031698
- [Background] Pogorelov P, Langenbucher A, Kruse F, Seitz B. Long-term results of phototherapeutic keratectomy for corneal map-dot-fingerprint dystrophy (Cogan-Guerry). Cornea. 2006 Aug;25(7):774-7. doi: 10.1097/01.ico.0000214801.02195.d4. PMID 17068452
- [Background] Gaster RN, Ben Margines J, Gaster DN, Li X, Rabinowitz YS. Comparison of the Effect of Epithelial Removal by Transepithelial Phototherapeutic Keratectomy or Manual Debridement on Cross-linking Procedures for Progressive Keratoconus. J Refract Surg. 2016 Oct 1;32(10):699-704. doi: 10.3928/1081597X-20160712-01. PMID 27722758
- [Background] Deshmukh R, Reddy JC, Rapuano CJ, Vaddavalli PK. Phototherapeutic keratectomy: Indications, methods and decision making. Indian J Ophthalmol. 2020 Dec;68(12):2856-2866. doi: 10.4103/ijo.IJO_1524_20. PMID 33229661
- [Background] Yeu E, Hashem O, Sheha H. Treatment of Epithelial Basement Membrane Dystrophy to Optimize the Ocular Surface Prior to Cataract Surgery. Clin Ophthalmol. 2022 Mar 15;16:785-795. doi: 10.2147/OPTH.S356421. eCollection 2022. PMID 35321046
- [Background] Buffault J, Zeboulon P, Liang H, Chiche A, Luzu J, Robin M, Rabut G, Labetoulle M, Labbe A, Baudouin C. Assessment of corneal epithelial thickness mapping in epithelial basement membrane dystrophy. PLoS One. 2020 Nov 25;15(11):e0239124. doi: 10.1371/journal.pone.0239124. eCollection 2020. PMID 33237913